CLINICAL TRIAL: NCT00998842
Title: Comparison of a Novel 12-Lead Wireless ECG and a Standard Wired ECG
Brief Title: Comparison of a Novel 12-Lead Wireless Electrocardiogram (ECG) and a Standard Wired ECG
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Thomas Allen, DO, University of Oklahoma
Other Study IDs: OU IRB 14853
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: ECG; EKG; healthy subjects; electrocardiography, ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- healthy subjects: five male, five female, ages 18-64
  Interventions: Device: Recom Model 100; Device: GE 5000 ECG Monitor System

INTERVENTIONS:
Device: Recom Model 100 — Battery Operated, Ambulatory, Digital Wireless ECG Monitor System
Device: GE 5000 ECG Monitor System — Wired ECG system

SUMMARY:
To determine if there is a difference between wireless ECG and wired ECG findings.

DETAILED DESCRIPTION:
The aim of the study is to compare ECG recordings from the Signalife Fidelity 100 Wireless 12-lead ECG Monitor System to that of the GE 5000 Wired 12-lead ECG Monitor System during rest and while walking. We hypothesize that ECG recordings from the wireless system will be equivalent to recordings from the standard wired system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals, AND
* Age 18-64

Exclusion Criteria:

* Pregnant women,
* Prisoners,
* Have known cardiovascular disease, OR
* Do not pass the PAR-Q and/or show baseline ECG abnormalities.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals Age 18-64
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
ECG recordings from the wireless system will be equivalent to recordings from the standard wired system. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Family Medicine Clinic, Tulsa, Oklahoma, United States